CLINICAL TRIAL: NCT03084887
Title: Intervention Study of Common Complications About Patients Placed Tissue Expansion Devices
Brief Title: Study of Tissue Expansion Devices Complications
Acronym: STEDC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KY20162083-1
Record Dates: First submitted 2017-02-04; First posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2016-11

CONDITIONS: Tissue Expansion
Keywords: Tissue Expansion Devices; Tissue Expansion; common complications; intervention study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- manuals and follow-up (Experimental): distribute manuals for patients before discharge and telephone follow-up per week until secondary hospital
  Interventions: Behavioral: manuals and follow-up
- controlled group (No Intervention): no intervention until secondary hospital

INTERVENTIONS:
Behavioral: manuals and follow-up — distribute manuals for patients before discharge and telephone follow-up per week until secondary hospital
  Arms: manuals and follow-up

SUMMARY:
Reduce the common complications incidence about patients placed tissue expansion devices to around 5%.

DETAILED DESCRIPTION:
Study design： Randomized parallel controlled trial. Study comments: 1.Telephone follow-up trainment group about 2-3 months until secondary hospital. 2.Promote the health management manual of patient placed expander,which includes discharge list, injection list, expander affusion operation procedure, injection myth, you ask me answer,injection record, injection diary record, appointment diaries etc.

ELIGIBILITY:
Inclusion Criteria:

* aged 1-70 years male and female;
* no complication when inclusion;
* sign the informed consent.

Exclusion Criteria:

* joined other clinical trial;
* occurred complications before inclusion;
* other infectious diseases;
* the pregnant or lactating women.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2016-11-10 (Actual); Primary Completion 2018-02-28 (Estimated); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
incidence of patients suffered the common complications | 2-3 months until secondary hospital
  count up the number of patients suffered the common complications

CONTACTS AND LOCATIONS:
Overall Officials: qing Yang, doctorate, Principal Investigator — First Affiliated Hospital of Fourth Military Medical University
Locations (1):
- xiaoling Wang, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided